CLINICAL TRIAL: NCT06375837
Title: Comparative Evaluation of an Alkasite-based Restorative Material and Two Different Resin Composites in Non-carious Cervical Lesions
Brief Title: Comparative Evaluation of an Alkasite-based Restorative Material and Two Different Resin Composites
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bioactive-NCCLs
Record Dates: First submitted 2023-10-02; First posted 2024-04-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Tooth Diseases
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- an alkasite-based restorative material (Experimental): Cention N, Ivoclar Vivadent, Schaan, Liechtenstein (CN) The liquid and powder will be mixed and then applied according to manufacturer's instructions.
  Interventions: Device: an alkasite-based restorative material
- hybrid resin composite (Experimental): Gradia Direct Anterior, GC, Tokyo, Japan (GR) After applying 37% orthophosphoric acid to the enamel of the lesions for 30 seconds and to the dentin for 15 seconds, the acid will be washed with water and then dried with light air. A universal adhesive (G-Premio Bond, GC, Tokyo, Japan) and then the composite will be applied according to the manufacturer's instructions.
  Interventions: Device: hybrid resin composite
- a highly filled flowable resin composite (Experimental): G-aenial Universal Flo, GC, Tokyo, Japan (GF) After applying 37% orthophosphoric acid to the enamel of the lesions for 30 seconds and to the dentin for 15 seconds, the acid will be washed with water and then dried with light air. A universal adhesive (G-Premio Bond, GC, Tokyo, Japan) and then the composite will be applied according to the manufacturer's instructions.
  Interventions: Device: a highly filled flowable resin composite

INTERVENTIONS:
Device: an alkasite-based restorative material — Cention N
  Arms: an alkasite-based restorative material
Device: hybrid resin composite — Gradia Direct Anterior
  Arms: hybrid resin composite
Device: a highly filled flowable resin composite — G-aenial Universal Flo
  Arms: a highly filled flowable resin composite

SUMMARY:
The clinical performance of an an alkasite-based restorative material and two different resin composites will be evaluated and compared in non-carious cervical lesions. After recruiting participants with at least three non-carious cervical lesions, all restorations will be placed by a single clinician. Lesions will be divided in three groups: an alkasite-based restorative material (Cention N, Ivoclar Vivadent, Schaan, Liechtenstein (CN)), hybrid resin composite (Gradia Direct Anterior, GC, Tokyo, Japan (GD)) and a highly filled flowable resin composite ((G-aenial Universal Flo, GC, Tokyo, Japan (GF)). All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using FDI criteria. Descriptive statistics will be performed using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* Age range will be 18 to 65.
* They will be required to have at least three NCCLs needed restoration in different teeth.
* All the NCCLs selected will be in similar sizes.

Exclusion Criteria:

* Patients with severe periodontal disease
* Patients with rampant, uncontrolled caries
* Patients with xerostomia
* Patients with serious medical problems preventing them from attending review visits
* Patients with poor gingival health
* Patients with heavy bruxism
* Patients with removable partial dentures
* Patients undergoing bleaching treatment or orthodontic treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different restorative systems according to FDI criteria (Esthetic properties) | two years
  Two year results according to FDI criteria. (Esthetic properties) The evaluations will be carried out using FDI criteria. Esthetic properties will be examined. Five scores will be given for each restoration: (1) Clinically excellent / very good, (2) Clinically good, (3) Clinically sufficient/satisfactory, (4) Clinically unsatisfactory, (5) Clinically poor.The data obtained for groups will be compared at each visit.

SECONDARY OUTCOMES:
Clinical performances of different restorative systems according to FDI criteria (Functional properties) | two years
  Two year results according to FDI criteria. (Functional properties) The evaluations will be carried out using FDI criteria. Functional properties will be examined.Five scores will be given for each restoration: (1) Clinically excellent / very good, (2) Clinically good, (3) Clinically sufficient/satisfactory, (4) Clinically unsatisfactory, (5) Clinically poor.The data obtained for groups will be compared at each visit.

OTHER OUTCOMES:
Clinical performances of different restorative systems according to FDI criteria (Biological properties) | two years
  Two year results according to FDI criteria. (Biological properties) The evaluations will be carried out using FDI criteria. Biological properties will be examined.Five scores will be given for each restoration: (1) Clinically excellent / very good, (2) Clinically good, (3) Clinically sufficient/satisfactory, (4) Clinically unsatisfactory, (5) Clinically poor.The data obtained for groups will be compared at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No